CLINICAL TRIAL: NCT02657460
Title: Clinical Trial of Tumor Cell-derived Microparticles Packaging Chemotherapeutic Drugs to Treat Malignant Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v1.4
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Malignant Pleural Effusion
Keywords: chemotherapy; microparticle; malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MTX-ATMPs (Experimental): methotrexate-autologous tumor derived microparticles
  Interventions: Biological: tumor derived microparticles
- cisplatin (Sham Comparator): Cisplatin is a traditional treatment for lung cancer
  Interventions: Drug: cisplatin

INTERVENTIONS:
Biological: tumor derived microparticles — The main difference between the two treatment groups is the biological coat, which is tumor derived microparticles.
  Arms: MTX-ATMPs
Drug: cisplatin — cisplatin is a traditional drug for lung cancer
  Other Names: cisplatinum
  Arms: cisplatin

SUMMARY:
The study is to investigate the anticancer effect and the related immunological mechanism of MTX-ATMPs in the treatment of malignant pleural effusion.

DETAILED DESCRIPTION:
Malignant pleural effusion(MPE) as a common complication of advanced lung cancer is lack of efficient treatments. The investigators have successfully produced tumor cell-derived microparticles packaging chemotherapy drugs and confirmed that this new integrative targeted biochemotherapy treatment could effectively restrain tumor growth at cellular and animal levels.This new method could control tumor growth in vivo effectively and induced pleural adhesion in the early clinical study. So the investigators attempt to explore the anticancer effect and related immune regulation mechanism of methotrexate-autologous tumor derived microparticles (MTX-ATMPs) in MPE treatment. The tumor cells in the malignant pleural effusion are prepared by screening, then MTX-ATMPs are made. Participants enrolled are randomly assigned to experimental and control group, each of them is injected with the prepared drug once in two days until the malignant pleural effusion are disappeared or the treatment cycle has been six times. During or after the whole treatment, reactions to each treatment of the participants are carefully followed up.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of lung cancer and malignant pleural effusion was confirmed by pathology and / or pleural fluid cytology;
2. The routine surgery or systemic radio/chemotherapy was ineffective, the MPE relapsed, or routine treatment therapy was given up by self-causes;
3. stable vital sign with KPS(Karnofsky Performance Status) index more than 60;
4. 18-70 years old;
5. normal haematopoietic function of bone marrow, no hemorrhagic tendency, blood routine test: HGB>=100g/L, WBC>4.0*10^9/L, PLT>80*10^9/L, serum ALT, AST within 2 times upper limit of normal, BUN within 1.5 time upper limit of normal, creatinine within normal range, normal EKG;
6. agreed to participate in the study and sign an informed consent;
7. without other severe comorbidities.

Exclusion Criteria:

1. lactating or pregnant patients;
2. allergy to multiple drugs;
3. with other severe comorbidities or psychological diseases;
4. severe infection;
5. participation in other clinical trials within the recent three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pleural effusions volume | four weeks

SECONDARY OUTCOMES:
Rivalta Test of pleural effusions | four weeks
total protein level of pleural effusions | four weeks
total karyocytes count of pleural effusions | four weeks
lactic dehydrogenase level of pleural effusions | four weeks
adenosine deaminase level of pleural effusions | four weeks
the cytology test of pleural effusions | four weeks
Karnofsky index | four weeks
survival time | six month
carcino embryonie antigen level in microgramme/L in serum | four weeks
CYFRA21-1 level in ng/mL in serum | four weeks
neuron specific annuals level in microgramme/L in serum | four weeks
squamous cell carcinoma antigen level in ng/mL in serum | four weeks
carcino embryonie antigen level in microgramme/L in pleural effusions | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jin, doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science & Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD now